CLINICAL TRIAL: NCT06657222
Title: A Multicenter FIH Dose Escalation and Optimization Phase I/IIa Trial to Investigate Safety, Tolerability, PK, and Efficacy of the 5T4 ADC TUB-030 in Patients With Advanced Solid Tumors (5-STAR 1-01)
Brief Title: First in Human Study of TUB-030 in Patients With Advanced Solid Tumors
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Tubulis GmbH (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: 5-STAR 1-01
Record Dates: First submitted 2024-10-15; First posted 2024-10-24 (Actual); Last update posted 2025-09-16 (Actual); Status verified 2025-09

CONDITIONS: Advanced Solid Tumors; HNSCC; SCLC; NSCLC; TNBC - Triple-Negative Breast Cancer; CRC
Keywords: Advanced Solid Tumors; NSCLC; Head and Neck Cancer
MeSH Terms: conditions — Squamous Cell Carcinoma of Head and Neck; Triple Negative Breast Neoplasms; Head and Neck Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Phase 1: dose escalation (Experimental): Drug TUB-030, administered by intravenous (IV) infusion
  Interventions: Drug: TUB-030
- Phase 2: dose optimization in NSCLC and HNSCC (Experimental): Drug TUB-030, administered by intravenous (IV) infusion NSCLC Cohort: Patients will be randomized to receive one of two doses administered by IV infusion HNSCC Cohort: Patients will be randomized to receive one of two doses administered by IV infusion
  Interventions: Drug: TUB-030

INTERVENTIONS:
Drug: TUB-030 — A complete treatment cycle is defined as 21 calendar days. TUB-030 will be administered as an intravenous (IV) solution on day 1 of each treatment cycle

SUMMARY:
The goal of this clinical trial is to learn if the drug TUB-030 works to treat solid cancer in adults. The study will also explore the safety of TUB-030. The main questions it aims to answer are:

To determine the safety and tolerability of TUB-030 To determine the maximum tolerated dose of TUB-030 as a single drug given to patients with solid cancer Researchers will also compare doses of TUB-030 in two specific cancer types, in patients with head and neck cancer and patients with non-small cell lung cancer, to see if TUB-030 works to treat these two solid cancer types and to determine the best dose.

Participants will:

Receive drug TUB-030 every 3 weeks Visit the clinic once every 3 weeks for checkups and tests Answer patient reported outcome questionnaires about their symptoms

ELIGIBILITY:
Inclusion Criteria:

1. Male or non-pregnant, non-breastfeeding female aged 18 years or older
2. Adequate organ function
3. Patients who received anti-cancer treatment including chemotherapy, biological therapy, endocrine therapy, PARP inhibitor, or other oral or investigational drugs must have had their last dose at least 4 weeks (6 weeks for nitrosourea, mitomycin-C) or 5 half-lives, whichever is shorter, before C1D1
4. AEs related to prior therapy, radiotherapy or surgical procedures must resolve to ≤grade 1.
5. For patients with known brain metastases, evidence of clinically stable disease post radiation therapy is required prior to enrollment.
6. For patients who underwent radiotherapy (≥ 30% of the bone marrow or wide field) to sites outside the brain, the final dose of radiation must have been administered ≥ 28 days prior to C1D1. For patients who underwent palliative radiotherapy (≤ 30% of the bone marrow or wide field) the final dose of radiation must have been administered ≥14 days prior to C1D1.
7. Radiologically measurable disease by RECIST v1.1, 4 weeks before C1D1, that can include a lesion in an irradiated field that shows progression according to RECIST v1.1 after irradiation.
8. Eastern Cooperative Oncology Group (ECOG) 0-1.
9. Have a life expectancy of >12 weeks for disease-related mortality, as evaluated by the INV.
10. In the opinion of the INV, the patient must be able and willing to understand and give signed informed consent
11. Women of childbearing potential (WOCBP) who are sexually active with a non-sterilized partner must use at least 1 highly effective method of contraception (with a failure rate of 1% per year) from the time of screening and must agree to continue using such precautions until the end of exposure, plus 5 half-lives and 6 months add-on in the case of patients of childbearing potential Patients must agree to continue a highly effective contraceptive method, refrain from egg cell donation and breastfeeding while on study treatment and for 5 half-lives plus 6 months after the last dose of study treatment.

Exclusion Criteria:

-

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 130 (Estimated)
Dates: Start 2024-12-13 (Actual); Primary Completion 2028-12 (Estimated); Study Completion 2028-12 (Estimated)

PRIMARY OUTCOMES:
Determination of MTD | From enrollment until 30 days after last study drug
  The highest dose is defined at which no more than 1 of 3 patients have had a Dose Limiting Toxicity (DLT) according to NCI CTCAE V5.0 criteria

SECONDARY OUTCOMES:
Number of patients with Adverse Events (AE) | From enrollment until 30 days after last study drug
  Any medical event in a participant which may or may not have a causal relationship with this treatment.
Maximum concentration (Cmax) | From enrollment until 30 days after last study drug
  The concentration of TUB-030 (conjugated ADC), total mAb, and free payload (Cmax will be derived).
Trough concentration (Cmin) | From enrollment until 30 days after last study drug
  The concentration of TUB-030 (conjugated ADC), total mAb, and free payload (Cmin will be derived).
The time taken to reach the maximum concentration (Tmax) | From enrollment until 30 days after last study drug
  The concentration of TUB-030 (conjugated ADC), total mAb, and free payload (Tmax will be derived).
Area Under Curve (AUC) | From enrollment until 30 days after last study drug
  PK endpoint
Half life (T1/2) | From enrollment until 30 days after last study drug
  PK endpoint
Determination of immunogenicity | From enrollment until 30 days after last study drug
  Number and percentage of patients developing anti-TUB-030 antibodies
Determination of efficacy | From enrolment until 30 days after last study drug.
  ORR by investigator assest Recist 1.1

CONTACTS AND LOCATIONS:
Overall Officials: Gunter Fingerle-Rowson, MD, PhD, Study Director — Tubulis GmbH
Locations (13):
- United States (12):
  - Yale Cancer Center, New Haven, Connecticut
  - University of Miami, Miami, Florida
  - Dana Farber Cancer Institute, Boston, Massachusetts
  - Mayo Clinic, Rochester, Minnesota
  - Washington University, St Louis, Missouri
  - Mount Sinai, New York, New York
  - Cleveland Clinic, Cleveland, Ohio
  - Ohio State University, Columbus, Ohio
  - NEXT Oncology Austin, Austin, Texas
  - NEXT Oncology - Dallas, Irving, Texas
  - NEXT Oncology - San Antonio, San Antonio, Texas
  - Fred Hutchinson Cancer Center, Seattle, Washington
- Princess Margaret, Toronto, Canada

IPD SHARING:
Plan to Share IPD: No
we first want to evaluate the ICMJE Guidelines